CLINICAL TRIAL: NCT06288685
Title: Percutaneous Trigger Finger Release Concomitant Steroid Injection Versus Percutaneous Trigger Finger Release Alone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Police General Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Weeraphat Saartying, Orthopedic Resident, Police General Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 73/256; 73/256 (Other: Police General Hospital)
Record Dates: First submitted 2024-02-17; First posted 2024-03-01 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Trigger Finger; Percutaneous A1 Pulley Release; Steroid Injection; Postoperative Pain
MeSH Terms: conditions — Trigger Finger Disorder; Pain, Postoperative | interventions — Triamcinolone

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with trigger finger, aged 18 years or older, and classified under Quinell's grade 2, 3, or 4, were included in the study [ ]. Recruitment took place at the Outpatient Orthopedic Department of the Police General Hospital between October 2023 and January 2024. Exclusion criteria encompassed individuals with a history of prior hand surgery, Dupuytren's disease, type 1 diabetes, previous phalangeal fractures, recent steroid injection within the last month, and autoimmune diseases.
Who Masked: Participant, Care Provider
Masking Description: Group allocation and Randomization:
  Patients were enrolled and randomized into two groups, percutaneous A1 pulley release with steroid injection (Group A) and percutaneous A1 pulley release alone (Group B), by utilizing computer generate randomization and the results were put in opaque sealed envelopes. Informed consent was obtained from all participants, and surgeries were performed by the same surgeon (WJ).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group1 (Experimental): percutaneous A1 pulley release with Triamcinolone injection
  Interventions: Procedure: percutaneous A1 pulley release; Drug: Triamcinolone
- group0 (Active Comparator): percutaneous A1 pulley release alone
  Interventions: Procedure: percutaneous A1 pulley release

INTERVENTIONS:
Procedure: percutaneous A1 pulley release — Treatment trigger finger by release A1 pulley by percutaneous procedure
Drug: Triamcinolone — Triamcinolone 40mg/ml 1 ml injection concomitant percutaneous A1 pulley release
  Arms: group1

SUMMARY:
Background:

Percutaneous A1 pulley release is a cost-effective and straightforward procedure with outcomes comparable to open A1 pulley release. Postoperative pain is a prevalent concern. Corticosteroid injection is a common nonoperative treatment for trigger finger, providing favorable outcomes but associated with a notable risk of recurrence. Numerous studies have explored the combined approach of percutaneous trigger finger release with corticosteroid injection. However, to date, there is no report on early postoperative results.

Objective:

To conduct a comparative analysis of early postoperative outcomes between percutaneous A1 pulley release with steroid injection and percutaneous A1 pulley release alone.

Study Design & Methods:

This study constitutes a randomized controlled trial involving patients with trigger finger who underwent percutaneous release surgery from October 2023 to January 2024. A total of 38 patients were enrolled, with 18 assigned to the percutaneous A1 pulley release with steroid injection group and 20 to the percutaneous A1 pulley release alone group. Postoperative assessments included pain scores using the Visual Analog Scale (VAS), evaluation of quality of life through the QuickDASH score (qDASH), patient satisfaction, and complications.

DETAILED DESCRIPTION:
Material and Methods

Study Population:

Patients diagnosed with trigger finger, aged 18 years or older, and classified under Quinell's grade 2, 3, or 4, were included in the study [ ]. Recruitment took place at the Outpatient Orthopedic Department of the Police General Hospital between October 2023 and January 2024. Exclusion criteria encompassed individuals with a history of prior hand surgery, Dupuytren's disease, type 1 diabetes, previous phalangeal fractures, recent steroid injection within the last month, and autoimmune diseases.

Group allocation and Randomization:

Patients were enrolled and randomized into two groups, percutaneous A1 pulley release with steroid injection (Group A) and percutaneous A1 pulley release alone (Group B), by utilizing computer generate randomization and the results were put in opaque sealed envelopes. Informed consent was obtained from all participants, and surgeries were performed by the same surgeon (WJ).

Surgical Technique:

The surgical procedure followed Eastwood's method [ ], involving the following steps:

1. Preparation of the sterile field.
2. Injection of 1% lidocaine with epinephrine at the surgical site.
3. Insertion of an 18-gauge needle following the tract from the previous injection.
4. Patient extension of the finger to bring flexor tendons close to the skin, moving the neurovascular structures away.
5. Slow penetration of the needle until it is over the A1 pulley.
6. Gentle flexion of the finger while observing the needle tip to prevent penetrating the flexor tendon.
7. Rotation of the needle bevel into a longitudinal orientation to the flexor tendon.
8. Release of the A1 pulley by moving the needle upward and downward parallel to the flexor tendon until complete release is achieved.
9. Withdrawal of the needle while hyperextending the finger.
10. Flexion and extension of the finger to check for triggering.
11. Injection of triamcinolone (40mg/ml) 1 ml in the study group.
12. Closure of the wound with a small elastic dressing.

Postoperative Protocols:

Both groups received identical postoperative protocols, including the same medications (Augmentin, Naproxen, Tolperisone) for 7 days. Patients were encouraged for early finger range of motion without restriction.

Outcome Measures:

The primary outcome measure was pain score assessed by the VAS. Secondary outcomes included quality of life measured by the qDASH score, patient satisfaction, and surgical complications.

Follow-Up:

All cases underwent follow-up via telephone on postoperative days 1 to 6, in the clinic during the first and second weeks, and at 1 to 2 months postoperative.

Statistical analysis In this study, all data calculations were conducted using Stata software (version 17.0). Group comparisons involved the application of Pearson's chi-squared test or Continuity Correction chi-squared test for categorical variables, and the student's t-test was employed for continuous variables. Statistically significant differences were defined as those with a P-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of trigger finger
* aged 18 years or older
* trigger finger are classified under Quinell's grade 2, 3, or 4

Exclusion Criteria:

* a history of prior hand surgery
* Dupuytren's disease
* type 1 diabetes
* previous phalangeal fractures
* recent steroid injection within the last month
* autoimmune diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain score | post operative Day0 until 2 months
  VAS(visual analog scale) from 0 to 10, 0 mean there is no pain, 10 there is the most pain in participants life

SECONDARY OUTCOMES:
hand function by quickDASH | post operative Day0 until 2 months
  quickDASH(questionnaire in Thai version), score from 0-100, 0 mean there is no limitation of daily hand activity, 100 mean participants got disability in that upper limb
patients satisfaction | post operative Day0 until 2 months
  1 is lowest satisfaction, 5 is most satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Police General Hospital, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Sharing the Dermographic data of the participants including age, BMI, Occupation and sharing of pain score, quality of life and satisfaction in result table
Supporting Information: Study Protocol, SAP, CSR
Time Frame: This may be from April 2024 until April 2029